CLINICAL TRIAL: NCT05305105
Title: Effects of Psilocybin in Post-Treatment Lyme Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Steven & Alexandra Cohen Foundation (Other); Usona Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00281685; 132642 (Other: Steven & Alexandra Cohen Foundation)
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Post-Treatment Lyme Disease; Chronic Lyme Disease; Lyme Disease, Chronic
Keywords: Psilocybin; Hallucinogen; Psychedelic
MeSH Terms: conditions — Post-Lyme Disease Syndrome | interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Psilocybin (Experimental): Participants will complete an 8-week course of study treatment including two doses of psilocybin with psychological support administered approximately 2 weeks apart.
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Dosing at the first session will be 15mg. For the second session participants will either remain at the initial dose, or increase to 25mg.

SUMMARY:
This study will examine the effects of psilocybin on Lyme disease symptom burden and quality of life in people with Post-Treatment Lyme Disease (PTLD).

DETAILED DESCRIPTION:
This pilot study will evaluate the therapeutic potential of psilocybin in people with well-documented current Post-Treatment Lyme Disease (PTLD). Study measures will assess the impact of psilocybin-assisted treatment on overall symptom burden and quality of life in 20 people with PTLD. This is an open-label proof-of-concept trial in which participants will complete an 8-week course of study treatment including two psilocybin sessions (15mg in week 4 and 15 or 25mg in week 6) with psychological support, and follow-up assessments 1, 3, and 6 months after the final psilocybin session.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age.
* Capable of providing written informed consent for participation into the study.
* Willingness to allow the study team to review past medical records.
* At least one current PTLD-defining symptom (widespread pain, fatigue, or neurocognitive dysfunction) following completion of standard, recommended antibiotic therapy for treatment of Lyme disease, and that appeared in the first two years following first evidence of Lyme disease.
* Medical record documentation of meeting the Centers for Disease Control (CDC) case definition for clear diagnosis and treatment of early or late Lyme disease while living in a Lyme-endemic area. In other words, a history of physician-documented single or disseminated erythema migrans rash, late Lyme arthritis, or late Lyme neuropathy, OR Medical record documentation of meeting the CDC case definition for probable early or late Lyme disease. In other words, a history of abrupt onset of flu-like symptoms with or without a misdiagnosed rash, and concurrent positive serology while living in a Lyme-endemic area.
* Received treatment with a recommended course of antibiotics.
* Be medically stable as determined by screening for medical problems via a personal interview, a medical questionnaire, a physical examination, an electrocardiogram (ECG), and routine medical blood and urinalysis laboratory tests.
* Concurrent pharmacotherapy with selective serotonin reuptake inhibitors (SSRI), serotonin and norepinephrine reuptake inhibitors (SNRI), and/or bupropion is allowed if the type and frequency of the therapy has been stable for at least two months prior to screening. Allowable bupropion doses for participants will be ≤300mg/day.

Exclusion Criteria:

* Meeting Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for moderate or severe substance use disorder (excluding tobacco) within the past 5 years.
* Currently taking antipsychotics, monoamine oxidase (MAO) inhibitors, or antidepressant medications other than SSRIs, SNRIs, or bupropion. Allowable bupropion doses for participants will be ≤300mg/day.
* Currently taking lithium or other primary centrally-acting serotonergic medications, whether over-the-counter or prescription (e.g., efavirenz, 5-hydroxytryptophan, St. John's wort).
* Cardiovascular conditions: angina, a clinically significant ECG abnormality (e.g. atrial fibrillation or corrected QT interval (QTc) >450msec), transient ischaemic attack (TIA) in the last 6 months, stroke, artificial heart valves, or uncontrolled hypertension with resting blood pressure systolic >139 or diastolic >89, or heart rate >90 bpm.
* Renal disease (creatinine clearance < 40 ml/min using the Cockcroft-Gault equation).
* Current or past history of meeting DSM-5 criteria for Schizophrenia, Psychotic Disorder (unless substance-induced or due to a medical condition), or Bipolar I or II Disorder.
* Family (i.e., 1st degree relative) history of Schizophrenia, Psychotic Disorder (unless substance-induced or due to a medical condition), or Bipolar I Disorder.
* Past-year hallucinogen use
* Received the Lyme vaccine when it was available (1998-2002).
* Development of unexplained chronic pain, chronic fatigue syndrome, fibromyalgia, autoimmune disease, or unexplained neurologic symptoms before first evidence of Lyme disease.
* Cancer or malignancy in the past 2 years.
* Epilepsy with history of seizures.
* Insulin-dependent diabetes; if taking oral hypoglycemic agent, then no history of hypoglycemia.
* Current dementia or related disorders including but not limited to, Alzheimer's Disease, vascular dementia, Lewy body dementia, and frontotemporal disorders.
* Current or past major immunosuppressive illness or medications.
* Currently pregnant or nursing.
* Currently of childbearing potential and not using effective methods of contraception.
* Not fluent in English.
* High risk for suicidal ideation or behavior (i.e., individuals who report suicidal ideation with intent or behavior on the Columbia-Suicide Severity Rating Scale (C-SSRS) at screening, or individuals with a suicide attempt within the past 3 years).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-10-26 (Actual); Study Completion 2025-04-07 (Actual)

PRIMARY OUTCOMES:
Change in multi-system symptom burden as assessed by the General Symptom Questionnaire (GSQ-30) score | Baseline, 2 weeks after final psilocybin dose, 1 month after final psilocybin dose
  The GSQ-30 is a validated and reliable instrument developed to assess multi-system symptom burden among patients with Lyme Disease. Total score ranges from 0 to 120, with higher scores indicating greater symptom burden.
Change in functional health and well-being as assessed by the Short Health Form (SF-36) score | Baseline, 2 weeks after final psilocybin dose, 1 month after final psilocybin dose
  The SF-36 (SF-36) is a multi-purpose, short form health survey that yields an 8-domain profile of functional health and well-being scores as well as psychometrically-based physical and mental health summary measures. The number of questions contributing to each domain varies from 2 to 10. Domain scores range from 0 (poorest health status) to 100 (best health status).

SECONDARY OUTCOMES:
Change in fatigue as assessed by the Fatigue Severity Scale (FSS) score | Baseline, 2 weeks after final psilocybin dose, 1 month after final psilocybin dose
  The FSS was designed to detect and evaluate changes in fatigue over time in persons with chronic illness. Its research utility rests with its ability to measure fatigue severity and identify features that distinguish fatigue between other clinical features of chronic medical disorders, such as depression. Scores on the FSS range from a minimum of 9 to a maximum of 63, with higher scores indicating greater fatigue severity.
Change in pain as assessed by the Short-Form McGill Pain Questionnaire (SF-MPQ) | Baseline, 2 weeks after final psilocybin dose, 1 month after final psilocybin dose
  The Short-Form McGill Pain Questionnaire (SF-MPQ) was designed to provide a quantitative measure of pain that can be tested statistically and includes major classes of word descriptors used by patients to specify subjective pain experience. The SF-MPQ 15-item pain metric has summary scores ranging from 0 to 45 with a higher score indicating worse pain.

OTHER OUTCOMES:
Change in depression as assessed by the Beck Depression Inventory-II (BDI-II) | Baseline, 2 weeks after final psilocybin dose, 1 month after final psilocybin dose
  The Beck Depression Inventory-II (BDI-II) is a widely used, validated, and reliable self-report instrument designed to assess the severity of depressive symptoms in adolescents and adults. Total score ranges from 0 to 63, with higher scores indicating greater depressive symptom severity.
Change in sleep quality as assessed by the Pittsburgh Sleep Quality Index (PSQI) | Baseline, 2 weeks after final psilocybin dose, 1 month after final psilocybin dose
  The Pittsburgh Sleep Quality Index (PSQI) is a validated and reliable instrument developed to assess subjective sleep quality and disturbances over a 1-month interval. Total score ranges from 0 to 21, with higher scores indicating poorer sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: Albert Garcia-Romeu, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fallon BA, Zubcevik N, Bennett C, Doshi S, Rebman AW, Kishon R, Moeller JR, Octavien NR, Aucott JN. The General Symptom Questionnaire-30 (GSQ-30): A Brief Measure of Multi-System Symptom Burden in Lyme Disease. Front Med (Lausanne). 2019 Dec 6;6:283. doi: 10.3389/fmed.2019.00283. eCollection 2019. PMID 31867334
- [Background] Rebman AW, Bechtold KT, Yang T, Mihm EA, Soloski MJ, Novak CB, Aucott JN. The Clinical, Symptom, and Quality-of-Life Characterization of a Well-Defined Group of Patients with Posttreatment Lyme Disease Syndrome. Front Med (Lausanne). 2017 Dec 14;4:224. doi: 10.3389/fmed.2017.00224. eCollection 2017. PMID 29312942
- See also: Online Study Screener — http://hopkinspsychedelic.org/lyme